CLINICAL TRIAL: NCT03604536
Title: Individualization of Oral Mesalazine Treatment Through a Self-managed Web-based Solution in Mild-to-moderate Ulcerative Colitis: A Pilot Study
Brief Title: Individualization Treatment Through a Self-managed Web-based Solution in Ulcerative Colitis
Status: Terminated | Type: Observational
Why Stopped: not able to recruit patients
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Petra Weimers, Prinicipal Investigator, Nordsjaellands Hospital
Other Study IDs: H-17038710
Record Dates: First submitted 2018-07-09; First posted 2018-07-27 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis
Keywords: Adherence; eHealth; Aminosalicylate
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study investigates the effect of individualized monotherapy with Mesalazine (Pentasa Sachet ®) on time to remission in patients with mild to moderate UC in an eHealth setting.

DETAILED DESCRIPTION:
More than 3 million Europeans suffer from inflammatory bowel disease (IBD), where Crohn's Disease (CD) and Ulcerative Colitis (UC) are the most common forms. They are chronic, relapsing and remitting diseases resulting in uncontrolled inflammation of the gastrointestinal (GI) tract with symptoms of diarrhoea, abdominal pain, weight loss and blood in the stools. The treatment aims to relieve and prevent GI tract inflammation and consists of anti-inflammatory and immunosuppressive drugs or surgical removal of the colon as a final option. The main treatment option for mild to moderate UC is Aminosalicylate. Mesalazine (5-aminosalicylic acid), both orally and topically, has been proven to be an effective treatment option for inducing as well as maintaining remission in patients with UC.

Pentasa Sachet are Mesalazine micro granules coated in ethyl cellulose with high (95%) 5-aminosalicylic acid (5-ASA) load. The coating provides a prolonged release of Mesalazine, allowing a continuous action from small bowel to rectum. Approximately 75% of the micro granules are released in the colon. This reduces the number of applications needed per day and is therefore considered to be a more desirable option by the patients. Once daily administrated 5-aminosalicylic acid (5-ASA) has been shown to be as effective as conventional dosing.

Fecal Calprotectin (FC) is an accurate biomarker of GI tract inflammation. FC correlates well with endoscopic disease activity and consequently serves as a substitute marker for mucosal healing as well as a clinical tool for disease monitoring. A home testing kit with a smart phone application, which only takes 18 min to carry out, has been developed. Thereby, facilitating the opportunity of telemonitoring of the disease course and stimulating patient engagement, empowerment and adherence to treatment.

Medication adherence is essential for maintaining remission, since non-adherence is one of the main causes of disease activity. A combined therapy of oral and topical 5-ASA is recommended by current guidelines for the treatment of active mild to moderate UC. However, patient adherence to oral 5-ASA is poor (approximately 60%), and even poorer to topical therapy (approximately 32%). A previous eHealth trial on individualized oral 5-ASA therapy reported higher adherence rates than previous studies on standard care. In addition, 90% of the study patients responded with remission on monotherapy and only 10% needed a combined therapy with topical treatment.

Web-based treating solutions (eHealth) have shown to optimize treatment effect in chronic diseases such as asthma, type 1 diabetes, and coagulation diseases. A web-based treatment solution for IBD patients, Constant-care, was in 1997 launched by Dr. Pia Munkholm. The web-program has since been proven to be an effective clinical tool, resulting in enhanced compliance, empowerment, improved quality of life and decreased relapse duration in IBD patients. Constant-Care consists of an education package and a disease-monitoring package. The disease monitoring part of the program is built upon an algorithm of two variables; FC and a validated disease activity questionnaire, Simple Clinical Colitis Activity Index (SCCAI) for UC patients. The FC values are acquired by the patients through a home testing kit and the disease activity questionnaire is filled out by the patients in the web- program. The eHealth system cumulates the data immediately, and subsequently presenting the result, a Total inflammatory Burden Score (TIBS), to the patients as a visual "traffic light" indicator of disease activity. Patients receive treatment advices by the program depending on the severity of the disease: green- remission, yellow- moderate activity, red-severe activity.

The disease monitoring part also consists of Patient-Related Outcome (PRO) questionnaires regarding quality of life, disability, fatigue, disease course type and compliance. The International Organization for the study of Inflammatory Bowel Disease (IOIBD) has since 2015 recommended the use of PRO's as a fundamental part of measuring treatment outcome in both UC and CD.

The primary aim of the study is to investigate the effect of individualized monotherapy with Mesalazine (Pentasa Sachet ®) on time to remission (clinical and Paraclinical (green TIBS)) in patients with mild to moderate UC in an eHealth setting. The investigators hypothesize that the web based therapy program will reduce the time to remission compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the Copenhagen Diagnostic criteria for UC
* Age between 18 and 75 years
* New and relapse patients diagnosed with Mild-to-moderate UC
* Current relapse (minimum 1 out of 2) SCCAI>2 (with a positive score in the variable of blood in stool) FC ≥200
* Diagnosed with left sided or extensive UC(24)
* Understand written and spoken Danish
* Easy access to internet and smartphone

Exclusion Criteria:

* Evidence of enteric infection
* Treatment with immunomodulators such as steroids, azathioprine, methotrexate, or infliximab within the last 8 weeks
* Two or more courses of oral steroids in the past 12 months
* Diagnosed with proctitis
* Severe disease activity (SCCAI >6 or FC ≥600)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with mild to moderate ulcerative colitis will be included from the Out patient clinic at the gastroenterology department, North Zealand University Hospital, Capitol region of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Total Inflammation Burden Scoring (TIBS) | At baseline and at 12 weeks or until remission, which ever comes first
  Self reported disease activity in combination with a fecal biomarker of inflammation (fecal calprotectin) results in TIBS. Disease activity is scored by 6 questions yielding: remission (<3) , mild to moderate disease activity (3-4) and severe disease activity ( >5). Fecal calprotectin: remission (<200mg/kg ), mild to moderate (200-599 mg/kg ), severe (>599 mg/kg). The two items are added together in a weighted manner giving the Total inflammation burden scoring (TIBS): remission (0-8), mild to moderate (9-32), severe (33-99).

SECONDARY OUTCOMES:
Disease course type | At baseline and after 12 weeks
  Self reported Disease course type according to the Copenhagen disease course type ( 5 different types). The five disease course types stretch from mild and indolent to constant active disease. In this study, patients have to choose one type representing their disease course since time of diagnosis, as well as at week 12 for the period since inclusion in the study.
Compliance with medication | at baseline and after 12 weeks
  self reported according to the Medicine Adherence Report Scale and visibility analog scale. Compliance scored according to Medicine Adherence Report Scale by 5 questions, and 1-5 points per question ( 5 = always, 1=never), maximum score 25. A score over 20 is considered god compliance.
  Visibility analog scale from 0-100, where 0 means no compliance and 100 means 100% compliant.
Short Inflammatory Bowel Disease Questionnaire | at baseline and after 12 weeks
  self reported quality of life according to the Short Inflammatory Bowel Disease Questionnaire, a disease specific health related quality of life questionnaire consisting of 10 questions in four domains: Emotional Health, Bowel Symptoms, Social Health and Work. The scoring range is from 10 (lowest score) to 70 (highest score). A cut-off level at >50 is interpreted as good health related quality of life.
Disability | at baseline and after 12 weeks
  self reported disability according to the IBD disk, consisting of 10 items: Abdominal pain, regulating defecation, interpersonal interactions, education and work, Sleep, energy, emotions, body image, sexual functions, joint pain. Patients can score from 0 (absolutely disagree/ no disability) to 10 (absolutely agree/severe disability) for each item. The results will be visualised to the patient as a coloured disc.
Fatigue | at baseline and after 12 weeks
  Fatigue is measured according to The Functional Assessment of Chronic Illness Therapy-Fatigue Scale, containing 13 questions to measure the fatigue component of health related quality of life. The scale ranges from 0-52 with zero being the worst possible score and 52 the best. A score of ≤30 represents fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Pia Munkholm, Prof, Study Director — North Zealand University Hospital
Locations (1):
- North zealand university hospital, Frederikssund, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinding KK, Elsberg H, Thorkilgaard T, Belard E, Pedersen N, Elkjaer M, Marker D, Carlsen K, Burisch J, Munkholm P. Fecal Calprotectin Measured By Patients at Home Using Smartphones--A New Clinical Tool in Monitoring Patients with Inflammatory Bowel Disease. Inflamm Bowel Dis. 2016 Feb;22(2):336-44. doi: 10.1097/MIB.0000000000000619. PMID 26535869
- [Background] Pedersen N, Thielsen P, Martinsen L, Bennedsen M, Haaber A, Langholz E, Vegh Z, Duricova D, Jess T, Bell S, Burisch J, Munkholm P. eHealth: individualization of mesalazine treatment through a self-managed web-based solution in mild-to-moderate ulcerative colitis. Inflamm Bowel Dis. 2014 Dec;20(12):2276-85. doi: 10.1097/MIB.0000000000000199. PMID 25248002
- [Background] Elkjaer M, Shuhaibar M, Burisch J, Bailey Y, Scherfig H, Laugesen B, Avnstrom S, Langholz E, O'Morain C, Lynge E, Munkholm P. E-health empowers patients with ulcerative colitis: a randomised controlled trial of the web-guided 'Constant-care' approach. Gut. 2010 Dec;59(12):1652-61. doi: 10.1136/gut.2010.220160. PMID 21071584
- [Background] Pedersen N, Elkjaer M, Duricova D, Burisch J, Dobrzanski C, Andersen NN, Jess T, Bendtsen F, Langholz E, Leotta S, Knudsen T, Thorsgaard N, Munkholm P. eHealth: individualisation of infliximab treatment and disease course via a self-managed web-based solution in Crohn's disease. Aliment Pharmacol Ther. 2012 Nov;36(9):840-9. doi: 10.1111/apt.12043. PMID 22971016